CLINICAL TRIAL: NCT02478294
Title: Evaluation of Thoracoscopic Left Atrial Appendage Excision Plus Atrial Fibrillation Ablation Versus Oral Anticoagulants for Secondary Prevention of Stroke and Non-central Nervous Systemic Embolism in Patients With AF: 5A Pilot Cohort
Brief Title: LAA Excision With AF Ablation Versus Oral Anticoagulants for Secondary Prevention of Stroke
Acronym: 5A
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Minglong Chen, Deputy Director of the Department of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2014-SR-113
Record Dates: First submitted 2015-06-12; First posted 2015-06-23 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation; Stroke; Systemic Embolism
Keywords: Atrial Fibrillation; Stroke; Systemic embolism; Left atrial appendage excision; Warfarin
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- the surgical intervention group: Thoracoscopic LAA Excision plus AF Ablation. Patients receiving thoracoscopic left atrial appendage excision plus atrial fibrillation alation
  Interventions: Procedure: Thoracoscopic LAA Excision plus AF Ablation
- oral anticoagulant treatment group: Warfarin or Novel Oral Anticoagulants. Patients receiving warfarin treatment (INR 2.0-3.0) or novel oral anticoagulants
  Interventions: Drug: Warfarin or Novel Oral Anticoagulants

INTERVENTIONS:
Procedure: Thoracoscopic LAA Excision plus AF Ablation — In this group, patients receive thoracoscopic LAA excision plus AF ablation, which means thoracoscopic left atrial appendage excision plus atrial fibrillation ablation.
  Groups: the surgical intervention group
Drug: Warfarin or Novel Oral Anticoagulants — In this group, patients receive warfarin or novel oral anticoagulants
  Groups: oral anticoagulant treatment group

SUMMARY:
This cohort study aims to evaluate thoracoscopic left atrial appendage excision plus atrial fibrillation ablation versus oral anticoagulants for the prevention of stroke and non-central nervous systemic embolism in patients with atrial fibrillation and thromboembolism.

DETAILED DESCRIPTION:
Brief Summary: This cohort study aims to compare thoracoscopic left atrial appendage excision plus atrial fibrillation ablation versus oral anticoagulants for secondary prevention of stroke and non-central nervous systemic embolism in patients with atrial fibrillation and thromboembolism.

Detailed Description: BACKGROUND: Atrial fibrillation (AF) is one of the most common cardiac arrhythmias and has been shown to be an important cause of stroke. AF is responsible for 15% of all strokes. Most strokes in AF are caused by cardioembolism. The left atrial appendage (LAA) is the dominant source of cardioembolism. The greatest priority in treating AF is stroke prevention. There are now 3 main approaches for prevention: (1) oral anticoagulation (OAC), (2) eradication of AF, and (3) exclusion of the LAA from the systemic circulation. OAC therapy, including warfarin and novel oral anticoagulants, effectively reduces the risk of stroke in AF and is currently the first line of treatment in patients with AF and one or more risk factors. Despite the advancements in medical therapy, the risk of stroke in patients with AF who undergo optimal anticoagulation therapy still remains between 2% and 5% per year, regardless of the agent used. The limitations of OAC include (1) patient unsuitability for OAC, (2) increased risk of bleeding, (3) need for monitoring optimal international normalized ratio (INR) levels (with warfarin), and (4) patient noncompliance. Percutaneous methods of ablation are widely used to attempt to eliminate AF. Approximately 20% of patients who underwent ablation had AF recurrence. It is because of this well-demonstrated occurrence that the guidelines do not recommend discontinuation of warfarin or equivalent therapies after ablation. Since at least 90% of all left atrial thrombi are found within the LAA, it is plausible that its occlusion will lead to a decreased risk of stroke in patients with AF. However, the evidence for surgical excision is extremely limited.

AIM OF THE STUDY: The primary objective of this study is to evaluate whether thoracoscopic LAA excision plus atrial fibrillation ablation for the purpose of prevention of thromboembolism in patients with AF and thromboembolism is more effective and safer compared with OACs for reducing the composite endpoint of stroke, TIA and systemic embolism. The primary end point was the composite of ischemic stroke/systemic embolism/transient ischemic attack (TIA), major bleeding, or all-cause mortality. The secondary end point is defined as ischemic strokes, all strokes (including ischemic and hemorrhagic), major and fatal bleeding events, minor bleeding complication, all-cause mortality, cardiovascular death, and hospitalization due to cardiovascular or cerebral diseases.

STUDY DESIGN: This is a single-center prospective cohort study. Adult patients with non-valvular AF and a previous history of ischemic stroke/systemic embolism/ TIA are eligible for inclusion of this study. Approximately 300 patients with paroxysmal or persistent AF and previous thromboembolic events will receive novel oral anticoagulant or warfarin treatment with a targeted INR between 2.0 and 3.0 or surgical LAA excision plus AF ablation. Follow-up for these patients includes visits at 3 m, 6 m, 9 m, 12 m, and every additional 6 months there after.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Have documented AF episodes
* The occurrence of ischemic stroke, TIA or systemic thromboembolism at least one month before enrollment
* Capable of understanding and signing the CRF

Exclusion Criteria:

* Reversible AF
* Modified Rankin score ≥4
* Having a history of rheumatic, severe valvular heart disease or heart valve replacement
* Having symptomatic carotid artery disease
* Having another disease which requires lifelong warfarin therapy
* Medical conditions limiting expected survival to <1 year
* Women of childbearing potential (unless post-menopausal or surgically sterile)
* Participation in any other clinical mortality trial
* Unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-valvular AF and a previous history of embolic events are eligible for inclusion of this study.
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
the composite of ischemic stroke/systemic embolism/transient ischemic attack (TIA), major bleeding, or all-cause mortality. | at least 3 month follow-up

SECONDARY OUTCOMES:
ischemic strokes | at least 3 month follow-up
all strokes (including ischemic and hemorrhagic) | at least 3 month follow-up
Major and fatal bleeding events | at least 3 month follow-up
Minor bleeding complication | at least 3 month follow-up
all-cause mortality | at least 3 month follow-up
cardiovascular death | at least 3 month follow-up
hospitalization due to cardiovascular or cerebral diseases | at least 3 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China